CLINICAL TRIAL: NCT05365373
Title: The Effect of Treatment Zone Decentration on Axial Length Elongation After Orthokeratology
Status: Completed | Type: Observational
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022005
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Myopia; Orthokeratology
Keywords: Myopia; Orthokeratology; Axial length; Decentration
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Orthokeratology lens is an effective method for myopia control. This study analyzed the effects of treatment zone decentration on axial length elongation in adolescents with orthokeratology lens.

DETAILED DESCRIPTION:
Orthokeratology lens is an effective method for myopia control. This study aimed to investigate the effects of treatment zone decentration on axial length elongation in adolescents with orthokeratology lens in 1 year. Other factors that may affect axial growth were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age from 8 to 15years
* spherical equivalent(SE) was range from -1.00D to -5.00D
* conform to the standard of wearing orthokeratology lens

Exclusion Criteria:

* ocular diseases and systemic diseases
* stop wearing for ≥7 days for any reason during the follow-up period
* keratoconjunctival complications, glare, diplopia, or any other symptoms during follow-up

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Myopia children with orthokeratology lens and complete follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The change of axial length | The change of baseline、6 months and 12months
  The axial length was measured by IOL-Master 500, its expressed in mm

SECONDARY OUTCOMES:
the decentration magnitudes of the treatment zone | up to 1 year
  The value of decentration magnitudes was obtained and calculated from a corneal topography

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No